CLINICAL TRIAL: NCT00360945
Title: Phase II Study of the Combination of Cisplatin + Temozolomide in Malignant Glial Tumours in Children and Adolescents at Diagnosis or in Relapse
Brief Title: Cisplatin and Temozolomide in Treating Young Patients With Malignant Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000482280; CCLG-CNS-2004-02; EU-20622
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2006-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood oligodendroglioma; untreated childhood cerebellar astrocytoma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Astrocytoma | interventions — Cisplatin; Temozolomide; In Situ Hybridization, Fluorescence; Immunohistochemistry; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: temozolomide
Genetic: fluorescence in situ hybridization
Genetic: loss of heterozygosity analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cisplatin together with temozolomide works in treating young patients with malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate (complete and partial response) in pediatric patients with malignant gliomas treated with temozolomide and cisplatin.

Secondary

* Identify genetic, metabolic, and proteomic profiles that will provide an insight into the molecular pathways involved in the pathogenesis of these tumors.
* Link genetic changes with clinical details, histopathology, and patient outcome, thereby developing a biological basis for diagnosis, prognosis, and treatment monitoring.
* Evaluate relapse-free survival at 1 and 2 years in patients treated at diagnosis.
* Evaluate the duration of clinical response in patients treated at relapse.
* Study the health status and quality of life of these patients.
* Evaluate long-term toxicity of this therapeutic combination.
* Evaluate the ability of magnetic resonance spectroscopy vs CT scan to predict response in patients with high-grade astrocytomas.

OUTLINE: This is a multicenter, open-label, nonrandomized, parallel-group study. Patients are stratified according to disease status (newly diagnosed vs relapsed). Patients with newly diagnosed disease are further stratified according to spread of disease (localized and measurable vs diffuse unmeasurable).

* Stratum I (newly diagnosed disease): Patients receive CISTEM chemotherapy comprising cisplatin IV over 3 hours on day 1 and oral temozolomide once daily on days 2-6. Treatment repeats every 28 days for up to 7 courses. Patients who achieve responsive or stable disease after 2 courses receive 2 more courses of CISTEM chemotherapy and then undergo radiotherapy 5 days a week for 6 weeks. After completion of radiotherapy, patients may receive up to 3 more courses of CISTEM chemotherapy for a total of 7 courses.
* Stratum II (relapsed disease): Patients receive CISTEM chemotherapy for up to 7 courses as in stratum I. Patients who reach the maximum dose allowed for cisplatin may receive oral temozolomide alone indefinitely.

Tissue and blood samples are obtained at baseline and examined by immunohistochemistry, fluorescent in situ hybridization (FISH), and loss of heterozygosity. The tumor tissue is analyzed for p53, MSH2, MLH1, and MGMT.

After completion of study treatment, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 87 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following grade III or grade IV malignant glial tumors*:

  * Glioblastoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic oligoastrocytoma
  * Anaplastic ganglioglioma
  * Anaplastic mixed tumor

    * Glial component is essential NOTE: *Malignant gliomas occurring as a second primary malignancy allowed
* Newly diagnosed or recurrent disease
* No malignant brain stem tumors
* Incompletely resected tumors

  * No completely resected tumors
* Measurable or evaluable disease by conventional MRI

PATIENT CHARACTERISTICS:

* Lansky performance status 40-100%
* Organ toxicity ≤ grade 2
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Prothrombin ≥ 50%
* Fibrinogen ≥ 1.5 g/L
* Creatinine normal for age

  * Creatinine ≤ 65 µmol/L (4-15 years of age)
  * Creatinine ≤ 110 µmol/L (15-20 years of age)
* Audiogram with toxicity grade ≤ 2
* ECG normal
* Negative pregnancy test
* Fertile patients must use effective contraception
* No severe or life-threatening infection
* No uncontrolled developing or symptomatic intracranial hypertension

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) or radiotherapy for patients with relapsed disease
* No prior cisplatin or temozolomide
* No other concurrent anticancer therapy

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Estimated)
Dates: Start 2004-04

PRIMARY OUTCOMES:
Response rate after 2 courses

SECONDARY OUTCOMES:
Relapse-free survival
Best response in patients receiving more than 2 courses
Rate of progression at 6 months and 1 and 2 years
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Steve Lowis, MD, PhD, BA, MRCP, MRCPCH — Bristol Royal Hospital for Children; Jacques Grill, MD, PhD — Gustave Roussy, Cancer Campus, Grand Paris; Anthony Michalski, MD — Great Ormond Street Hospital for Children NHS Foundation Trust; David A. Walker — Queen's Medical Center
Locations (23):
- Institut Gustave Roussy, Villejuif, France
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (21):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Middlesex Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton University Hospital NHS Trust, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales